CLINICAL TRIAL: NCT05153395
Title: Novel Treatment for Brain Insulin Resistance and Hypoperfusion
Brief Title: Impact of Intranasal Insulin on Sympathetic Activity and Cerebral Vasodilation
Status: Suspended | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Interim data and power analysis
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Jacqueline K Limberg, PhD, Associate Professor, University of Missouri-Columbia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2057288
Record Dates: First submitted 2021-11-18; First posted 2021-12-10 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Healthy; Vasodilation; Insulin Resistance; Autonomic Dysfunction; Obesity
MeSH Terms: conditions — Aneurysm; Insulin Resistance; Primary Dysautonomias; Obesity | interventions — Neurovascular Coupling; Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Insulin (Doppler) (Experimental): Human insulin (160 IU) will be administered as a bolus using an intra-nasal device.
  Interventions: Other: Carbon dioxide breathing; Other: Neurovascular Coupling; Drug: Human insulin
- Insulin (MRI) (Experimental): Human insulin (160 IU) will be administered as a bolus using an intra-nasal device.
  Interventions: Other: Carbon dioxide breathing; Drug: Human insulin
- Time Control (Doppler) (Other): Time control only
  Interventions: Other: Carbon dioxide breathing; Other: Neurovascular Coupling

INTERVENTIONS:
Other: Carbon dioxide breathing — Hypercapnic (5% carbon dioxide) air will be administered before and after intra-nasal insulin exposure.
Other: Neurovascular Coupling — Participants will be asked to repeatedly open and close their eyes. With eyes open, participants will focus on a visual image. This will be done before and after intra-nasal insulin exposure.
  Arms: Insulin (Doppler); Time Control (Doppler)
Drug: Human insulin — Participants will be administered human insulin (160 IU) as a bolus using an intra-nasal device.
  Arms: Insulin (Doppler); Insulin (MRI)

SUMMARY:
The purpose of this project is to examine the impact of increases in brain insulin on sympathetic nervous system activity, as well as peripheral and cerebral blood flow in humans.

ELIGIBILITY:
Inclusion Criteria:

* healthy adult men and women;
* 18-45 years of age;
* BMI >18 kg/m2;
* non-pregnant/non-breastfeeding;
* non-nicotine users;

Exclusion Criteria:

* taking any medications known to affect metabolic, respiratory, cardiovascular, and/or autonomic

Self-reported history of:

* hepatic, renal, pulmonary, cardiovascular, or neurological disease;
* stroke or neurovascular disease;
* bleeding/clotting disorders;
* sleep apnea or other sleep disorders;
* diabetes;
* smoking;
* history of alcoholism or substance abuse;
* hypertension;
* respiratory disease;
* active cancer;
* autoimmune disease.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 65 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Amount of cerebral blood flow | Change from baseline at minute 15
  Measured with trans-cranial Doppler ultrasound (cm/s) or arterial spin labeling (mL/100 g/min)

SECONDARY OUTCOMES:
Amount of muscle sympathetic nerve activity (MSNA) | Change from baseline at minute 15
  MSNA burst incidence (bursts/100 heart beats)
Amount of leg blood flow | Change from baseline at minute 15
  Measured with Doppler ultrasound (mL/min)

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline K Limberg, Ph.D., Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided